CLINICAL TRIAL: NCT02585141
Title: Aspiration or Surgical Drainage of Perianal Abscess. A Randomized Controlled Clinical Study
Brief Title: Aspiration Treatment of Perianal Abscess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Karam Matlub Sørensen, Principal Investigator, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-20140191
Record Dates: First submitted 2015-10-15; First posted 2015-10-23 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Anal Fistulas
MeSH Terms: conditions — Rectal Fistula | interventions — Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- aspiration (Experimental): Aspiration of perianal abscess(MEDIPLAST® 13 G, 2,5 x 110 mm) under general anesthesia followed by antibiotic treatment with Clindamycin tablet 300 mg 3 times daily for 7 days
  Interventions: Device: MEDIPLAST® (aspiration); Drug: Clindamycin
- incision (Active Comparator): Surgical incision of perianal abscess under general anesthesia.
  Interventions: Procedure: incision

INTERVENTIONS:
Device: MEDIPLAST® (aspiration) — The aspiration drainage will be with a large caliber needle (MEDIPLAST® 13 G, 2,5 x 110 mm) and a syringe of 20 ml. The cavity must be emptied for pus and irrigated by repeated injection and aspiration of saline until clear fluid is obtained.
  Arms: aspiration
Procedure: incision — Incision drainage will be undertaken as standardized de-roofing of the abscess and debridement. Wound packing and dressing will not be used, just sitz bath or ordinary hygiene until wound healing.
  Arms: incision
Drug: Clindamycin — Postoperative broad spectrum oral antibiotics covering both aerobes and anaerobes bacteria will be given for seven days of Clindamycin 300 mg tablets x 3 a day
  Other Names: postoperative antibiotic
  Arms: aspiration

SUMMARY:
The purpose of this study is to compare aspiration and oral antibiotics with surgical incision in the treatment of perianal abscesses in terms of recurrence and subsequent fistula formation. Included patients will be randomised to either aspiration or incision.

DETAILED DESCRIPTION:
Anorectal abscess is a common condition, caused by cryptoglandular polymicrobial infection, where the traditional treatment is surgical drainage. Anorectal abscess is associated with recurrence rates between 6-44 % after surgical drainage and persistent subsequent fistula up to 37 %. Inadequate incision, missed abscess components or fistulas can be the cause of recurrence . Surgical drainage is associated with discomfort from prolonged wound healing, affecting the daily activities as well as the potential risk of complicated scaring and fecal incontinence. Less invasive method with pus aspiration under antibiotic cover has been shown to be safe in terms of recurrence rate and subsequent fistula formation and well tolerated by the patients with less morbidity and wound complications and a potential lower risk of fecal incontinence. However, this has been shown only in few studies with small population and no randomized controlled study comparing the two approaches has been conducted or published to our knowledge. The risk factors of recurrence and subsequent fistula formation are not that clear but age below 40 years, absence of diabetes mellitus and recent smoking are shown to be risk factors for developing recurrent abscess and fistula. Applying aspiration and antibiotics method for the treatment of perianal abscess can be an advantage for the society due to a shorter recovering period, quicker return to daily activity and work and avoiding wound healing problems and sphincter damage; thus lower expenses. The results of this study have the potentials to reveal the risk factors of developing fistula after perianal abscess.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 yrs old
2. Perianal abscess (without spontaneous rupture)
3. Abscess larger than 2 cm in diameter
4. Signed informed consent

Exclusion Criteria:

1. Malignancy within 5 yrs
2. Previous radiotherapy of the abdomen and pelvis
3. Recurrent abscess within 6 months
4. Immune suppressed patients
5. Pregnant and lactating women
6. Abscess with horseshoe formation
7. Allergy to Clindamycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in recurrence rate | 2,12 and 52 weeks
  Rate of recurrences of abscesses in each arm after 2,12 and 52 weeks

SECONDARY OUTCOMES:
changes in Quality of life score | 2,12 and 52 weeks
  Changes in Short Form Health Survey (SF-36) questionaire after 2,12 and 52 weeks
fecal incontinence | 2,12 and 52 weeks
  changes in Wexner fecal incontinence score after 2,12 and 52 weeks
Risk factors for fistula formation and abscess recurrence | 2,12 and 52 weeks
  risk factors for recurrences and fistula formation as; age, gender, BMI, smoking and alcohol use. Furthermore presence or absence of the following medical conditions: diabetes mellitus, ischemic cardiac disease, arrhythmia, hypertension, asthma/ COLD, connective tissue disease and renal function impairment. As well as the characteristics of perianal abscess: number of abscesses, localization, distance from anus in cm, largest diameter in cm, length of symptoms and use of antibiotics prior to admission. Finally bacterial culture.Risk factors of developing fistula after both treatments; both medical and abscess related will be analyzed using multivariate analysis.
Changes in healing time | 2,12 and 52 weeks
  time to recovery and wound healing after both procedures and it will be measured as the number of days between operation and healed wound.
Changes in fistulas formation | 2,12 and 52 weeks
  rate of fistula formation in each arm after 2,12 and 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Karam M Sørensen, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Background] Marcus RH, Stine RJ, Cohen MA. Perirectal abscess. Ann Emerg Med. 1995 May;25(5):597-603. doi: 10.1016/s0196-0644(95)70170-2. PMID 7741334
- [Background] Hamalainen KP, Sainio AP. Incidence of fistulas after drainage of acute anorectal abscesses. Dis Colon Rectum. 1998 Nov;41(11):1357-61; discussion 1361-2. doi: 10.1007/BF02237048. PMID 9823799
- [Background] Kovalcik PJ, Peniston RL, Cross GH. Anorectal abscess. Surg Gynecol Obstet. 1979 Dec;149(6):884-6. PMID 505265
- [Background] Read DR, Abcarian H. A prospective survey of 474 patients with anorectal abscess. Dis Colon Rectum. 1979 Nov-Dec;22(8):566-8. doi: 10.1007/BF02587008. PMID 527452
- [Background] Vasilevsky CA, Gordon PH. The incidence of recurrent abscesses or fistula-in-ano following anorectal suppuration. Dis Colon Rectum. 1984 Feb;27(2):126-30. doi: 10.1007/BF02553995. PMID 6697831
- [Background] Cox SW, Senagore AJ, Luchtefeld MA, Mazier WP. Outcome after incision and drainage with fistulotomy for ischiorectal abscess. Am Surg. 1997 Aug;63(8):686-9. PMID 9247434
- [Background] Chrabot CM, Prasad ML, Abcarian H. Recurrent anorectal abscesses. Dis Colon Rectum. 1983 Feb;26(2):105-8. doi: 10.1007/BF02562586. PMID 6822168
- [Background] Malik AI, Nelson RL, Tou S. Incision and drainage of perianal abscess with or without treatment of anal fistula. Cochrane Database Syst Rev. 2010 Jul 7;(7):CD006827. doi: 10.1002/14651858.CD006827.pub2. PMID 20614450
- [Background] Rickard MJ. Anal abscesses and fistulas. ANZ J Surg. 2005 Jan-Feb;75(1-2):64-72. doi: 10.1111/j.1445-2197.2005.03280.x. PMID 15740520
- [Background] Beck DE, Fazio VW, Lavery IC, Jagelman DG, Weakley FL. Catheter drainage of ischiorectal abscesses. South Med J. 1988 Apr;81(4):444-6. doi: 10.1097/00007611-198804000-00008. PMID 3358166
- [Background] Kyle S, Isbister WH. Management of anorectal abscesses: comparison between traditional incision and packing and de Pezzer catheter drainage. Aust N Z J Surg. 1990 Feb;60(2):129-31. PMID 2327914
- [Background] Kronborg O, Olsen H. Incision and drainage v. incision, curettage and suture under antibiotic cover in anorectal abscess. A randomized study with 3-year follow-up. Acta Chir Scand. 1984;150(8):689-92. PMID 6397949
- [Background] Isbister WH. A simple method for the management of anorectal abscess. Aust N Z J Surg. 1987 Oct;57(10):771-4. doi: 10.1111/j.1445-2197.1987.tb01259.x. PMID 3426451
- [Background] Mortensen J, Kraglund K, Klaerke M, Jaeger G, Svane S, Bone J. Primary suture of anorectal abscess. A randomized study comparing treatment with clindamycin vs. clindamycin and Gentacoll. Dis Colon Rectum. 1995 Apr;38(4):398-401. doi: 10.1007/BF02054229. PMID 7720448
- [Background] Lohsiriwat V, Yodying H, Lohsiriwat D. Incidence and factors influencing the development of fistula-in-ano after incision and drainage of perianal abscesses. J Med Assoc Thai. 2010 Jan;93(1):61-5. PMID 20196412
- [Background] Devaraj B, Khabassi S, Cosman BC. Recent smoking is a risk factor for anal abscess and fistula. Dis Colon Rectum. 2011 Jun;54(6):681-5. doi: 10.1007/DCR.0b013e31820e7c7a. PMID 21552051
- [Background] Hamadani A, Haigh PI, Liu IL, Abbas MA. Who is at risk for developing chronic anal fistula or recurrent anal sepsis after initial perianal abscess? Dis Colon Rectum. 2009 Feb;52(2):217-21. doi: 10.1007/DCR.0b013e31819a5c52. PMID 19279415
- [Background] Smieja M. Current indications for the use of clindamycin: A critical review. Can J Infect Dis. 1998 Jan;9(1):22-8. doi: 10.1155/1998/538090. PMID 22346533
- [Background] Stevens DL, Bisno AL, Chambers HF, Everett ED, Dellinger P, Goldstein EJ, Gorbach SL, Hirschmann JV, Kaplan EL, Montoya JG, Wade JC; Infectious Diseases Society of America. Practice guidelines for the diagnosis and management of skin and soft-tissue infections. Clin Infect Dis. 2005 Nov 15;41(10):1373-406. doi: 10.1086/497143. Epub 2005 Oct 14. No abstract available. PMID 16231249
- [Derived] Sorensen KM, Moller S, Qvist N. Needle aspiration treatment vs. incision of acute simple perianal abscess: randomized controlled study. Int J Colorectal Dis. 2021 Mar;36(3):581-588. doi: 10.1007/s00384-021-03845-6. Epub 2021 Jan 15. PMID 33447866
- See also: OPEN homepage. OPEN hosts all projects data. — http://open.rsyd.dk/OpenProjects/da/openProject.jsp?openNo=145